CLINICAL TRIAL: NCT01272739
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of IHBG-10 on Weight Loss and Body Composition
Brief Title: Randomized Study to Evaluate the Effect of an Investigational Product on Weight Loss and Body Composition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI-1300-IHBG10
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-01

CONDITIONS: Obesity
Keywords: obesity; weight loss; weight management; overweight; nutriceutical
MeSH Terms: conditions — Obesity; Weight Loss; Overweight | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Experimental): Subjects will take 500 mg of the investigational product 15 minutes prior to the 3 main meals of the day.
  Interventions: Dietary Supplement: IHBG-10
- Control Group (Placebo Comparator): Subjects will take a placebo 15 minutes prior to the three main meals of the day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IHBG-10 — 500 mg of IHBG-10 taken 15 minutes prior to the three main meals of the day
  Other Names: IHBG10
  Arms: Study Group
Dietary Supplement: Placebo — Placebo taken 15 minutes prior to the three main meals of the day
  Other Names: sugar pill
  Arms: Control Group

SUMMARY:
This is a pilot study to determine the safety and efficacy of an investigational product (IHBG-10) on weight loss, and changes in body composition.

DETAILED DESCRIPTION:
Subjects will be randomized to one of two groups: one group will take 500 mg of the investigational product (IHBG-10) 15 minutes prior to the three main meals of the day; the other group will take placebo 15 minutes prior to the three main meals of the day. Subjects will be on the investigational product or placebo for 12 weeks. Participation in this study involves four study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Body mass index of 30 or greater
* Agree to keep diet, exercise and all current health habits stable during participation in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding or planning to become pregnant
* Prior bariatric surgery
* Use of prescription or over-the-counter appetite suppressants, herbal products or other medications for weight loss within the past month
* Obesity as a result of a clinically diagnosed endocrine problem
* Currently taking an anti-psychotic medication
* History of peptic ulcer disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Weight | 12 weeks

SECONDARY OUTCOMES:
Body composition | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward Zawada, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States